CLINICAL TRIAL: NCT00693576
Title: The Effect of Simvastatin on Desensitization of Panel-Positive Kidney Transplant Candidates
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Shiraz university of medical science, Shiraz university of medical science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2519
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Renal Transplantation
Keywords: renal transplant; panel reactive antibody; sensitization; simvastatin; immunological
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): patients who will take simvastatin 20 mg daily
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — 20 mg simvastatin daily

SUMMARY:
Patients with panel reactive antibodies have many difficulties to find a crossmatch-negative kidney for transplantation and are at the risk of post transplantation rejection more than other transplanted patients. We evaluated the effect of simvastatin on PRA and post transplant outcome of these sensitized patients. We also performed a descriptive study.

DETAILED DESCRIPTION:
The presence of panel reactive antibodies (PRAs) in the sera of renal transplant candidates is associated with hyperacute or delayed humoral immune responses against the graft after transplantation .

In addition, these sensitized patients wait for a long time to find a cross-match negative kidney for renal transplantation . As a result, some modalities have been used for desensitization including plasmapheresis and intravenous immunoglobulin (IVIG) in combination with immunosuppressive drugs .

However, recently, the use of statins such as simvastatin, pravastatin and etc. has been proposed to be safer and more effective for desensitization .

ELIGIBILITY:
Inclusion Criteria:

1. patients with ESRD on hemodialysis or peritoneal dialysis
2. On the waiting list for renal transplant
3. PRA more than 25%

Exclusion Criteria:

1. Pregnant women
2. Patients who need ongoing blood products
3. Patients taking other therapies to decrease PRA
4. Patients listed for multi-organ transplant other than kidney
5. Patients with liver failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
effect of simvastatin on panel reactive antibody | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: jamshid roozbeh, associate professor, Study Director — shiraz university of medical science; azar Sattarinezhad, internal medicine resident, Principal Investigator — shiraz university of medical science,internal medicine department; mohammad mahdi sagheb, assistant professor, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran